CLINICAL TRIAL: NCT05563727
Title: Prospective Evaluation of Sedation-related Complications During Gastroenterological Procedures
Brief Title: Sedation-related Complications During Gastroenterological Procedures
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Selin Erel, Attending Anesthesiologist in Gazi University School of Medicine, Gazi University
Other Study IDs: 238(23.12.2021)
Record Dates: First submitted 2022-08-29; First posted 2022-10-03 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Complication of Anesthesia; Sedation-related Complications
Keywords: sedation; gastroenterolojical procedure; complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Applications of non-operating room anesthesia for diagnosis and treatment are required in a variety of disciplines nowadays. Although it is not painful, sedation may be required in the gastrointestinal unit during procedures that put the patient through discomfort and stress, in order to reduce anxiety and provide analgesia. The purpose of this study is to evaluate the sedation used in our hospital's gastrointestinal endoscopy unit in light of intraoperative hemodynamic variables and perioperative problems. There are studies about non-operating room anesthesia in the literature, but there aren't many of them in our country, and none of them include a number of participants. The size of this study will exceed any study in Turkey.

DETAILED DESCRIPTION:
All patients will be informed about the study before the gastroenterological procedure and the consent form will be signed by the patients who want to participate in the study. Demographic data of patients (age, weight, height), ASA (American Society of Anesthesiologists) classification, allergies, comorbidities (hypertension, coronary artery disease, chronic kidney disease, COPD), Mallampati scores, history of covid, history of covid vaccine, and history of previous anesthesia will be questioned and recorded before the gastroenterological procedure. Afterward, participants will be taken to the gastroenterology intervention room and standard monitorisation (Electrocardiogram, noninvasive blood pressure, peripheral oxygen saturation, and end-tidal CO2) will be performed. The measurements will be repeated every 5 minutes following the induction of anesthesia and recorded. Administered anesthetics and their doses at the induction and maintenance of sedation will be recorded. The person recording the data will not be the patient's primary anesthesiologist. The data will be recorded by a second anesthesiologist who will not interfere with the medical treatment and management of the patient. The presence of perioperative and postoperative complications (such as hypotension, hypertension, bradycardia, apnea, hypoxia, agitation, postoperative nausea and vomiting) will be observed by the second anesthesiologist and recorded. Hypertension is defined as an elevation in blood pressure more than 20% compared to perioperative values. Hypotension is defined as degradation in blood pressure more than 20% compared to perioperative values. Bradycardia is defined as less than 50 heartbeats per minute. Peripheral oxygen saturation below 90 will be referred to as hypoxia. Apnea is defined as "no respiratory effort for more than 20 seconds" or "a halt of breathing for more than 10 seconds. There will be no intervention for the patients. Patients will not be divided into groups or randomized. The data will be recorded by an impartial observer.

ELIGIBILITY:
Inclusion Criteria:

* All patients who agree to participate in the study will be included
* Patients who will be sedated for an elective procedure in gastroenterology

Exclusion Criteria:

* pediatric patients (<18 years)
* who did not want to participate in the study
* mentally retarded patients
* language problems (not knowing turkish)
* emergent interventions
* allergy to the anesthetics
* need for endotracheal intubation or general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients participating in the study will be required to sign a voluntary consent form.
  Patients who will undergo gastroenterological intervention (such as will be included.
  endoscopy, colonoscopy, endocolon, endoscopic ultrasonography, endoscopic submucosal dissection, endoscopic retrograde cholangiopancreatography) in a single central gastroenterology intervention unit in our hospital.
Sampling Method: Probability Sample
Enrollment: 693 (Actual)
Dates: Start 2021-12-25 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
The relationship between different anesthetic drugs and complications will be investigated | 8 months
  During gastroenterological procedures, drugs such as propofol, ketamine, fentanyl, lidocaine, and midazolam are used in different combinations. Which anesthetic medicines induce complications like hypertension, hypotension, hypoxia, apnea, bradycardia, nausea, vomiting, and agitation to be more noticeable will be investigated in our study. Hypertension is defined as an elevation in blood pressure more than 20% compared to perioperative values. Hypotension is defined as degradation in blood pressure more than 20% compared to perioperative values. Bradycardia is defined as less than 50 heartbeats per minute. Peripheral oxygen saturation below 90 will be referred to as hypoxia. Apnea is defined as "no respiratory effort for more than 20 seconds" or "a halt of breathing for more than 10 seconds. For statistical analyses, a binomial logistic regression model will be established to determine the risk factors for complications according to drug type and complications.
The relationship between comorbidities and complications | 8 months
  Patients who will undergo a gastroenterological procedure may have different comorbidities such as hypertension, chronic arterial disease, diabetes, COPD, and chronic kidney disease. We want to investigate which comorbidities are more likely to result in particular complications in our study. For statistical analyses, a binomial logistic regression model will be established to determine the risk factors for complications according to comorbidities.

SECONDARY OUTCOMES:
Incidence of sedation related complications in gastroenterology unit | 8 months
  All the complications will be recorded and the most common ones will be revealed.

CONTACTS AND LOCATIONS:
Overall Officials: Selin Erel, Principal Investigator — Gazi Üniversitesi Tıp Fakültesi
Locations (1):
- Gazi University School of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After the data is collected and statistically analyzed, the study will be shared with the literature as an article
Supporting Information: Study Protocol, CSR
Time Frame: 1 year